CLINICAL TRIAL: NCT01388647
Title: Phase I/II Study of Neoadjuvant Carboplatin, Eribulin Mesylate and Trastuzumab (ECH) for Operable HER2 Positive Breast Cancer
Brief Title: Study of Neoadjuvant Carboplatin, Eribulin and Trastuzumab for Operable HER2 Positive Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closed early due to increased hematologic toxicity and possible reduced efficacy
Sponsor: Vector Oncology (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALSSNBC1006
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Results first posted 2015-08-28 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2014-12

CONDITIONS: HER-2 Positive Breast Cancer
Keywords: Neoadjuvant Treatment; HER-2 Positive Breast Cancer
MeSH Terms: interventions — eribulin; Carboplatin; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eribulin, carboplatin, and trastuzumab (Experimental): During Phase I, the eribulin dose will be assigned upon study enrollment. The maximum tolerated dose (MTD) determined in Phase I will be the dose used for Phase II. Eribulin will be administered intravenously (IV) over 2 to 5 minutes on Days 1 and 8 of each cycle. Carboplatin area under the curve (AUC) 6 will be administered IV over 15 to 30 minutes on Day 1 of each cycle. Trastuzumab will be administered as an IV infusion on Day 1 of each cycle. A loading dose of 8 mg/kg of trastuzumab will be administered over 90 minutes on Cycle 1 Day 1. Then, a maintenance dose of 6 mg/kg of trastuzumab will be administered over 30 to 90 minutes on Day 1 of Cycles 2 - 6.
  Interventions: Drug: eribulin; Drug: carboplatin; Drug: trastuzumab

INTERVENTIONS:
Drug: eribulin — During Phase I, the eribulin dose will be assigned upon study enrollment. The maximum tolerated dose (MTD) determined in Phase I will be the dose used for Phase II. Eribulin will be administered intravenously (IV) over 2 to 5 minutes on Days 1 and 8 of each cycle.
  Other Names: eribulin mesylate; HALAVEN
Drug: carboplatin — Carboplatin area under the curve (AUC) 6 will be administered IV over 15 to 30 minutes on Day 1 of each cycle.
Drug: trastuzumab — Trastuzumab will be administered as an IV infusion on Day 1 of each cycle. A loading dose of 8 mg/kg of trastuzumab will be administered over 90 minutes on Cycle 1 Day 1. Then, a maintenance dose of 6 mg/kg of trastuzumab will be administered over 30 to 90 minutes on Day 1 of Cycles 2 - 6.
  Other Names: Herceptin

SUMMARY:
This study will evaluate the safety and efficacy of eribulin in combination with carboplatin and trastuzumab in the neoadjuvant setting in subjects who are human epidermal growth factor receptor (HER)2 positive and are clinically stage IIA to IIIB.

The study regimen will be administered every 3 weeks for a total of 6 cycles followed by definitive surgery.

DETAILED DESCRIPTION:
During Phase I, the eribulin dose will be assigned upon study enrollment. The maximum tolerated dose (MTD) determined in Phase I will be the dose used for Phase II. Eribulin will be administered intravenously (IV) over 2 to 5 minutes on Days 1 and 8 of each cycle. Carboplatin area under the curve (AUC) 6 will be administered IV over 15 to 30 minutes on Day 1 of each cycle. Trastuzumab will be administered as an IV infusion on Day 1 of each cycle. A loading dose of 8 mg/kg of trastuzumab will be administered over 90 minutes on Cycle 1 Day 1. Then, a maintenance dose of 6 mg/kg of trastuzumab will be administered over 30 to 90 minutes on Day 1 of Cycles 2 - 6.

eribulin: During Phase I, the eribulin dose will be assigned upon study enrollment. The maximum tolerated dose (MTD) determined in Phase I will be the dose used for Phase II. Eribulin will be administered intravenously (IV) over 2 to 5 minutes on Days 1 and 8 of each cycle.

carboplatin: Carboplatin area under the curve

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Females; 18 years of age or greater
* Histologically proven invasive breast cancer
* American Joint Committee on Cancer (AJCC) clinical stage IIA - IIIB
* Tumor size greater than 10 millimeters
* HER2 positive
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Estrogen receptor (ER) positive or negative
* Ejection fraction greater than or equal to lower limit of normal for the institution by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA)
* Less than or equal to Grade 1 neuropathy according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
* Planned lumpectomy or mastectomy
* Eligible for radiation therapy
* No prior treatment for invasive breast cancer
* Adequate organ system function per protocol as determined within 7 days prior to first dose of study treatment
* Women of childbearing potential must have a negative pregnancy test within 7 days prior to the first dose of study treatment and must agree to use adequate contraception methods during study treatment and for a minimum of 6 months following trastuzumab discontinuation
* Female subjects who are lactating should discontinue nursing prior to the first dose of study treatment and should refrain from nursing throughout the treatment period

Exclusion Criteria:

* Fine needle cytology only without other histologic evidence of invasive breast cancer
* Inflammatory breast cancer
* AJCC clinical stage T1a-b breast cancer (primary tumor less than or equal to 10 millimeters)
* Evidence of metastatic disease
* HER2 negative
* Ejection fraction less than lower limit of normal for the institution by ECHO or MUGA
* Corrected QT interval greater than 480 milliseconds
* Pre-existing cardiac dysfunction
* Prior history of invasive cancer within the past 3 years
* Synchronous bilateral breast cancer
* Pre-existing CTCAE v4.0 Grade 2 or greater neuropathy
* Hypersensitivity to halichondrin B or halichondrin B chemical derivative
* History of severe allergic reactions to cisplatin or other platinum containing compounds, or mannitol
* Mild, moderate, or severe hepatic impairment
* Moderate or severe renal impairment
* Hypokalemia or hypomagnesemia if it cannot be corrected prior to the first dose of study treatment
* Organ allografts requiring immunosuppression
* Known positive human immunodeficiency virus (HIV) status
* Prior major surgery within 28 days prior to the first dose of study treatment and/or presence of any non-healing wound, fracture, or ulcer
* Minor surgery or radiation therapy within 14 days prior to the first dose of study treatment
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Schwartzberg, MD, FACP, Study Chair — Vector Oncology and The West Clinic
Locations (4):
- United States (4):
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Northeast Georgia Cancer Care, Athens, Georgia
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - The West Clinic, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to enrollment at four community oncology centers in the United States from July 2011 to June 2014.
Pre-assignment Details: Informed consent was obtained from all subjects. Subjects must have had no prior treatment for invasive breast cancer.
Groups:
- Eribulin 1.1 mg/m2: Subjects assigned to receive a starting dose of eribulin 1.1 mg/m2
- Eribulin 1.4 mg/m2: Subjects assigned to receive a starting dose of eribulin 1.4 mg/m2
Period: Overall Study
Arm/Group | Eribulin 1.1 mg/m2 | Eribulin 1.4 mg/m2
Started | 6 | 6
Completed | 5 (one subject ended study treatment due to adverse events) | 4 (two subjects ended study treatment due to adverse events)
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eribulin 1.1 mg/m2 | Eribulin 1.4 mg/m2 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (7.47) | 53.0 (9.14) | 53.1 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.4 (6.79) | 32.4 (4.59) | 32.4 (5.52)

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Response
Description: Definitive surgery will be performed 3 to 8 weeks after completion of study treatment. The pathology report will be scored for pathologic response: complete pathologic response (no invasive cancer in breast or lymph nodes; residual DCIS or LCIS is acceptable), partial pathologic response (residual invasive cancer in breast and/or lymph nodes), or no response (pathologic staging is equal to or worse than pretreatment clinical staging).
Time Frame: Assessed at time of definitive surgery, approximately 21-26 weeks from study treatment start
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eribulin 1.1 mg/m2 | Eribulin 1.4 mg/m2
Number analyzed (Participants) | 6 | 6
percentage of participants
  Complete Response | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1]
  Partial Response | 83.3 [35.9 to 99.6] | 83.3 [35.9 to 99.6]

2. Secondary Outcome: Clinical Response
Description: Clinical assessment of response will be performed 3 weeks after completion of study treatment. The treating physician will assess clinical response using physical examination and radiologic evaluation. Clinical response options are complete response (no invasive tumor in breast and lymph nodes), partial response (> 50% reduction in longest diameter of pretreatment tumor), no response (< 50% response to 10% growth of tumor as determined by longest diameter of pretreatment tumor size), and progression.
Time Frame: Assessed prior to definitive surgery, approximately 18 weeks from study treatment start.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eribulin 1.1 mg/m2 | Eribulin 1.4 mg/m2
Number analyzed (Participants) | 6 | 6
percentage of participants
  Complete Response | 16.7 [0.4 to 64.1] | 50.0 [11.8 to 88.2]
  Partial Response | 83.3 [35.9 to 99.6] | 33.3 [4.3 to 77.7]
  Missing | 0 [0 to 0] | 16.7 [0.4 to 64.1]

3. Other Pre Specified Outcome: Maximum Tolerated Dose (MTD) of Eribulin in Combination With Carboplatin and Trastuzuamb
Description: The MTD is defined as the dose at which <= 1 of 6 subjects experience DLT (Dose Limiting Toxicity) and above which >= 2 of 6 subjects experience DLT.
Time Frame: Approximately 22 days from study treatment start, per subject
Population: The MTD of ECH as neoadjuvant therapy for HER2+ breast cancer was determined per protocol definitions; however, due to the combination of increased hematologic toxicity and possible reduced efficacy, Phase II of this trial was not initiated.
Measure: Number; unit: mg/m^2
Groups:
- All Study Participants: All subjects were assigned to receive either a starting dose of eribulin 1.1 mg/m^2 or eribulin 1.4 mg/m^2.
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
mg/m^2 | 1.1

4. Other Pre Specified Outcome: Dose Limiting Toxicity (DLT)
Description: DLT is defined as grade 4 thrombocytopenia; grade 4 anemia; grade 4 neutropenia lasting > 5 days; or any grade 3 or 4 non-hematologic toxicity occurring during Cycle 1 which is attributable to eribulin, carboplatin, trastuzumab or the combination, or the inability to deliver all three agents at the assigned dose and scheduled time during Cycle 1.The following events are excluded from the DLT definition: grade 3 nausea and/or vomiting responsive to antiemetics; grade 3 fever or infection; grade 3 diarrhea responsive to antidiarrheal therapy.
Time Frame: Approximately 22 days from study treatment start, per subject
Measure: Number; unit: participants
Arm/Group | Eribulin 1.1 mg/m2 | Eribulin 1.4 mg/m2
Number analyzed (Participants) | 6 | 6
participants
  Grade 4 thrombocytopenia | 1 | 1
  Inability to deliver all 3 agents at assigned dose | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning at the start of study treatment until 21 days after the subject's last study treatment
Arm/Group | Eribulin 1.1 mg/m2 | Eribulin 1.4 mg/m2
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin 1.1 mg/m2 (N=6) | Eribulin 1.4 mg/m2 (N=6)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Aortitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin 1.1 mg/m2 (N=6) | Eribulin 1.4 mg/m2 (N=6)
Anemia (Blood and lymphatic system disorders) | 5 | 3
Iron Deficiency Anemia (Blood and lymphatic system disorders) | 1 | 1
Hypophosphatasia (Congenital, familial and genetic disorders) | 0 | 1
Hearing Impaired (Ear and labyrinth disorders) | 0 | 1
Vision Blurred (Eye disorders) | 1 | 1
Abdominal Distension (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 4 | 6
Vomiting (Gastrointestinal disorders) | 2 | 4
Adverse Drug Reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 2
Fatigue (General disorders) | 5 | 4
Gait Disturbance (General disorders) | 0 | 2
Mucosal Inflammation (General disorders) | 0 | 1
Edema Peripheral (General disorders) | 1 | 2
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 3
Hypersensitivity (Immune system disorders) | 2 | 0
Seasonal Allergy (Immune system disorders) | 0 | 1
Skin Infection (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 2
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 4 | 5
Occult Blood Positive (Investigations) | 0 | 1
Platelet Count Decreased (Investigations) | 5 | 3
Romberg Test Positive (Investigations) | 0 | 1
Weight Decreased (Investigations) | 0 | 1
White Blood Cell Count Decreased (Investigations) | 2 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 4
Hypouricemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Ataxia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 3
Dysgeusia (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 3 | 3
Hypoesthesia (Nervous system disorders) | 0 | 1
Hyporeflexia (Nervous system disorders) | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 3
Syncope (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Breast Discharge (Reproductive system and breast disorders) | 1 | 0
Breast Pain (Reproductive system and breast disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Antibiotic Prophylasis (Surgical and medical procedures) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Lymphedema (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Although MTD of eribulin with carboplatin & trastuzuamb as neoadjuvant therapy was determined by protocol definitions, study closed early due to increased hematologic toxicity & possible reduced efficacy. Phase II of this trial was not initiated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less